CLINICAL TRIAL: NCT04716985
Title: Evaluation of the Daily Intake of 0.5 L of Water Saturated With Molecular Hydrogen for 21 Days in COVID-19 Patients Treated in Ambulatory Care. Double-blind, Randomized, Comparative Study
Brief Title: Evaluation of the Daily Intake of 0.5 L of Water Saturated With Molecular Hydrogen for 21 Days in COVID-19 Patients Treated in Ambulatory Care
Acronym: HYDRO COVID
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: AGIR à Dom (Other)
Collaborators: Laboratoire TIMC-IMAG (Other); DrinkHRW, British Columbia, Canada (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2020-A03137-32
Record Dates: First submitted 2021-01-13; First posted 2021-01-20 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: SARS-CoV-2; Covid19; AMBULATORY CARE
Keywords: MOLECULAR HYDROGEN; anti-inflammatory role
MeSH Terms: conditions — COVID-19 | interventions — Hydrogen

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, multicentre comparative study.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: They will be labeled study (randomization number to respect blind and legal notices labeling clinical research).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TREATMENT GROUP (Active Comparator): Water saturated with molecular hydrogen at the rate of 2 times 250 mL / day for 21 days.
  80 mg of Mg metal, and safe excipients (dextrose, malic acid, L-tartaric acid, adipic acid).
  Interventions: Dietary Supplement: MOLECULAR HYDROGEN
- PLACEBO GROUP (Placebo Comparator): Water saturated with magnesium at the rate of 2 times 250 mL / day for 21 days. 80 mg of Mg, but in ionic form.
  Interventions: Dietary Supplement: PLACEBO MAGNESIUM

INTERVENTIONS:
Dietary Supplement: MOLECULAR HYDROGEN — Magnesium Tablet
  Arms: TREATMENT GROUP
Dietary Supplement: PLACEBO MAGNESIUM — Magnesium carbonate tablet
  Arms: PLACEBO GROUP

SUMMARY:
Through its anti-inflammatory role, molecular hydrogen could have a beneficial effect in preventing the runaway inflammatory reactions that lead to complications of Covid-19.

This hypothesis is supported by numerous preclinical and theoretical arguments, as well as by some Chinese clinical studies (the Chinese guidelines for the management of Covid-19 recommend the inhalation of hydrogen), a recommendation whose interest has just been confirmed by a publication describing the very positive results of a clinical study in China.

Through its anti-inflammatory role, molecular hydrogen could have a beneficial effect in preventing the runaway inflammatory reactions that lead to complications of Covid-19.

The ingestion of water saturated with molecular hydrogen has been the subject of several clinical studies in other indications than Covid-19, and no side effects of this ingestion have been reported. A recent publication recommends initiating clinical trials using a hydrogen fortified beverage.

DETAILED DESCRIPTION:
CURRENT STATE OF KNOWLEDGE ON PATHOLOGY :

SARS-CoV-2 is the causative agent of a new infectious respiratory disease called Covid-19 (for CoronaVirus Disease 2019) which is characterized primarily by potentially serious and fatal lung damage. The seriousness of the clinical signs associated with this pathology requires hospital admission of approximately 20% of patients, of which 5 to 10% will be admitted to intensive care. The more severe forms, though seen mainly in people over 60 years old, also occur in younger patients, most of whom are affected by comorbidities such as hypertension (30%), diabetes (17 %) or cardiovascular pathologies (15%). The mortality due to this infection varies according to the series between 2 and 14%. The most severe cases of this pathology begin with dyspnea which rapidly worsens around the 7th to 10th day of the disease into Acute Respiratory Distress Syndrome (ARDS) which requires the patient to be mechanically ventilated in the intensive care unit. and is responsible for the majority of deaths. ARDS is an active feature of severe forms of Sars-Cov-2 infection, directly linked to the mortality of this infection. The clinico-radiological aspect is not specific to other aetiologies of ARDS. Certain biological parameters suggest a massive and sudden release of cytokines (interleukins IL-6, IL-8 and IL-10 mainly) secondary to a syndrome of macrophage activation mainly at the pulmonary level. This cytokine storm is comparable to that of secondary hemophagocytic lymphohistiocytosis which occurs in approximately 4% of sepsis and is accompanied, in 50% of cases, by ARDS. The effect of this inflammatory cascade leads to an uncontrolled influx and activation of polynuclear and macrophagic cells with hyperproduction of oxygen-derived free radicals. These reactive species will damage the capillary alveolar membrane with initially hyperpermeability, and secondarily with fibrosis and fibroblast proliferation.

Several therapeutic trials aimed at reducing or controlling this immune storm are underway (anti-IL-6 antibodies, anti-r IL6 antibodies, corticosteroids).

PROPOSED STRATEGY, PURPOSE AND NOVELTY OF THE STUDY :

There are many theoretical, preclinical and clinical arguments to suggest that the administration of molecular hydrogen (H2) could, by the original anti-inflammatory effect of H2, help to avoid the cytokine storm. These arguments justified the launch of clinical trials proposing the inhalation of H2 (the investigators submitted to the French Ministry of Health (ANSM) a protocol, which has just been accepted by the ANSM, providing for the inhalation of H2 in patients Covid-19 at the start of oxygen therapy). As will be described in the next section, inhalation delivers significantly more H2 than ingestion of water saturated with H2. However, the inhalation of H2 involves a complex intervention, which in practice can only be considered late, as it can only be implemented for the benefit of hospitalized patients, typically in addition to oxygen therapy.

However, the arguments in favor of the potential interest of H2 in preventing the consequences of the cytokine storm apply particularly at the very beginning of the pathology: it would be very useful to be able to prevent not the consequences, but the occurrence of this storm, which would imply a very early intervention. It is this thinking that motivates this clinical trial.

The investigators hypothesis is that the early ingestion of water enriched in H2, through its anti-inflammatory effect, could prevent the complications of Covid-19 in the short, medium and long term. The investigators have found no evidence of any clinical study proposing to explore this original route, which does not use a drug, but a product classified and marketed as a dietary supplement.

To be able to demonstrate this effect, it is preferable to address a population in which the prevalence of complications is high. The investigators have therefore chosen to target patients over the age of 60 or 18 to 59 years old with at least one risk factor, in whom the complication rate is of the order of 50%. To explore the effect of a very early administration of H2, the investigators will limit themselves to patients at the very beginning of the pathology, symptomatic for no more than 5 days with the realization of a nasopharyngeal sample for COVID- 19, or asymptomatic contact subjects diagnosed with COVID + by RT-PCR or antigen test, the contagion dating no more than 10 days, and who may remain at home, without treatment or with routine care not requiring oxygen therapy. The patients in the interventional arm will self-administer H2, by ingesting 2 x 250 mL for 21 days, i.e. 0.5 L of water enriched in H2 per day, which they will manufacture themselves by dissolving 80 mg tablets of Mg metal (supplied by DrinkHRW, British Columbia, Canada): this was the method which seemed to us to be the simplest and easiest to implement for self-administration at home. Patients in the control group will receive an effervescent placebo tablet containing the same dose of Mg, but in ionic form, unable to generate H2 on contact with water.

The primary endpoint will be a composite endpoint combining worsening of symptoms (dyspnea and fatigue), putting on 02, hospitalizations and death occurring within 12 to 14 days following a PCR COVID-19 + diagnosis.

CURRENT KNOWLEDGE ON THE EXPLORATIONS PROVIDED FOR BY THE PROTOCOL :

Molecular hydrogen (H2) acts on the final path of the complex inflammatory cascade leading to the cytokine storm, by inhibiting the cellular action of reactive oxygen species.

Although the first study on the protective effects of hydrogen reported in the literature dates back to the 1970s, it is an experimental study on the therapeutic effects of molecular hydrogen in a model of cerebral infarction in rats which really constituted the starting point for numerous experimental works in animals and humans. This study showed that hydrogen enrichment (2-4%) of inspired air significantly decreases the volume of necrosis resulting from experimental cerebral ischemia in rats. The authors' interpretation was that the protective effect of molecular hydrogen was due to an antioxidant action linked to its reducing properties and its ability to diffuse easily through cell membranes. However, other studies quickly showed that the antioxidant and anti-free radical properties of hydrogen alone are not sufficient to explain the anti-inflammatory and anti-apoptotic effects of hydrogen administration. Thus, a study have shown that hydrogen inhibits the intracellular signaling pathways of inflammation without involving anti-free radical effects.

In addition, inhalation of hydrogen (2.9%) also limits the activation of mast cells. Finally, a study showed that two 60-minute sessions of inhalation of a gas mixture containing 2% hydrogen made it possible to limit lesions and mortality of multiple organs in a model of generalized inflammation in mice. The same authors have shown that inhalation of hydrogen restores the PaO2 / FiO2 ratio, both in a mouse model of sepsis by cecal ligation and in a model of lung disease induced by lipopolysaccharides (LPS). In view of the current data in the literature, the application of a treatment with molecular hydrogen makes it possible to trigger many potentially protective mechanisms in a hyperinflammatory context, such as sepsis and very probably Covid-19, by trapping hydroxyl radicals and peroxynitrite, by limiting inflammatory reactions by modulating intracellular transduction cascades and by modifying the expression of certain genes. This has been confirmed and specified in the case of Covid-19 by a very recent publication.

Several routes of administration have been used for hydrogen, they have been widely implemented in the clinic. The most widely used today, both in animals and in clinical trials in humans, are the ingestion of drinking water enriched in hydrogen and the inhalation of a gas mixture containing up to 4% of hydrogen. The inhalation route allows for the administration of much larger amounts of H2 than ingestion of H2 enriched water. In fact, as Ohta reports, inhalation makes it possible to permanently maintain a high concentration of H2 in the liquid compartments, whereas, less than an hour after ingestion of water enriched in H2, the concentration in the organism of molecular hydrogen returns to its baseline.

The preparation of water enriched with H2 can be done in several ways, and consumers have access to it in the context of "general public" products, excluding health products, considered as well-being products or as food supplements. Multiple CE marked water electrolysis devices are available on the French market, they can easily be implemented at home by interested consumers (see for example http://www.alkavoda.com/product/hydrogen- water-generator / or https://www.lifeionizers.com/products/alkaline-water-ionizers/). Hydrogenated water can also be produced industrially by electrolysis, and distributed in the form of flexible aluminum bags (see for example https://susosuwater.com/products/packages). Finally, the consumer can produce his hydrogenated water himself, by dissolving a tablet of magnesium metal in a cup (see for example https://drinkhrw.com/, which will provide us with the 80 mg tablets of Mg metal). Mg metal reacts spontaneously with water, according to the reaction Mg + 2H20 -> Mg (OH) 2 + H2. This last approach allows to have a hydrogen supersaturation for about 10 minutes, then the H2 concentration returns to the saturation limit (800 micromoles / L), with a half-life of one hour thereafter. The investigators will therefore recommend that the patient dissolve one Mg tablet in 250 mL of water twice a day, to drink as much water as possible (ideally at least 200 mL) immediately after dissolving this tablet (approximately 90 mL/s), and the rest as soon as possible, while remaining within the limits of an ingestion deemed comfortable by the patient.

No side effects of the administration of H2 could be demonstrated by the numerous preclinical and clinical studies. Some studies have even been carried out with high pressure gas mixtures (60 bars) containing 49% H2, which corresponds to a considerably greater administration of H2 than inhalation of mixtures with 4% H2 at atmospheric pressure, and therefore even more than what can be administered by ingestion (this was during deep diving experiments, the mixture was used to prevent decompression sickness and arterial thrombi. There are traces at https://clinicaltrials.gov/ of 20 clinical trials involving inhalation or ingestion of hydrogen, but there are more globally, as research in this area is much more active in Japan , not all of the trials of which are listed on this site, and more recently in China, where two trials on the benefit of inhalation of H2 in Covid-19 by an original method have been launched, one of which is still in progress. A first publication highlights the protective effect against the complications of Covid by inhaling a mixture containing 66% H2. Regarding the ingestion of water enriched in H2, Ohta lists numerous clinical trials. The investigators carried out a literature review themselves, which found a total of 410 patients included in clinical trials involving the ingestion of water enriched in H2. Among the recent trials whose methodology is similar to that which the investigators are considering, the investigators note a Japanese double-blind randomized trial including 178 patients with Parkinson's disease, patients in the interventional arm received 1 L of H2-saturated water for 48 weeks: no side effects has been noted. Finally, note the recent mini-review which concludes that the ingestion of water supersaturated with H2 (and also containing citrulline) is of potential interest in COVID-19.

Finally, it should be noted that the FDA has published a note classifying hydrogen-enriched water as GRAS (Generally Regarded As Safe), see http://www.rexresearch.com/bghealth/ucm409796.pdf and more specifically published a note accepting the tablets designed by DrinkHRW as "New Dietary Ingredient", specifying the conditions of use that the investigators will implement in this project.

Since the discovery of the first cases of Covid-19 in China, different strategies have been adopted to contain the inflammatory response of patients through antioxidant approaches. In this context, at least three pilot studies [https://www.cebm.net/covid-19/registered-trials-and-analysis/] and one multicenter clinical study [https://clinicaltrials.gov/ct2/show / NCT04336462? Cond = hydrogen + covid + 19 & draw = 2 & rank = 1] have been launched in China since January 2020, using the reducing properties of molecular hydrogen. The first results of these studies have been very encouraging, to such an extent that the Chinese health authorities have included hydrogen therapy in the guidelines on the management of patients hospitalized with moderate Covid-19 [Diagnosis and Treatment Protocol for Novel Coronavirus Pneumonia (Trial Version 7), National Health Commission & State Administration of Traditional Chinese Medicine. March 3, 2020].

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 59 years old or over 60 years old.
* If patient 18 to 59 years old, presence of at least one risk factor :

  * Hypertension under treatment (all stages)
  * Obesity (BMI ≥30 kg / m2)
  * Diabetes under treatment (all types)
  * Stable ischemic heart disease (all stages)
  * Atrial fibrillation
  * Stable heart failure (all stages)
  * History of stroke
  * Stage 3 chronic renal failure (30 ≤ estimated GFR <60 mL / min / 1.73 m²)
  * COPD (all stages, including chronic respiratory failure under long-term oxygen therapy)
  * Solid tumors or malignant hemopathies that are progressive or whose diagnosis is less than 5 years old
  * Immunodeficiency:
* of therapeutic origin (solid organ transplantation or transplant of hematopoietic stem cells, anticancer chemotherapy, immunosuppressive treatment, corticosteroid therapy> 15 mg / day equivalent to prednisone price for at least 2 months);
* or HIV infection and last known CD4 count <200 / mm3

  * History of pulmonary embolism and / or proximal deep vein thrombosis
  * Asthma under inhaled corticosteroid therapy
  * Paired sleep apnea syndrome
  * Peripheral arterial disease of the lower limbs stage II and above
  * Another risk factor presented, according to the list defined by the French High Council of Public Health
  * OR Presence of at least 3 comorbidities, according to the Rapid Responses to COVID-19 from the French High Council of Public Health.
* Patient with nasopharyngeal swab (antigenic test, RT-PCR, or other HAS-validated swabs to come) :

  * In case of positive test (antigenic test, RT-PCR, Other), patient with at least 1 symptom at the time of testing:
  * In case of negative antigenic or other test or ongoing or uninterpretable RT-PCR test, the patient must present at least 3 of the 11 symptoms of COVID-19 dating back no more than 4 days as defined below and notion of contact (with a certain or probable COVID+ patient) dating back less than 10 days:

Fever > 37,5°C since 3 days Cough Sore throat/cold Headache Anosmia, dysgeusia Myalgias, arthralgias, bone pain Respiratory difficulties (feeling of dyspnea at rest) Chest pain (sternal) Digestive complaints (diarrhea, nausea, vomiting) Tachycardia (palpitation) Conjunctivitis (red eyes)

* No seriousness signs during the consultation and for at least 72 hours.
* Patient able to understand the procedure and follow it and have tools for a video-consultation.
* Affiliation to the social security system.
* Voluntary to participate to the study, informed consent form signed after appropriate information

Exclusion Criteria:

* The absence of attending or referring physician
* Any sign of seriousness incompatible with home care.
* Severe chronic kidney failure or dialysis (i.e. DFGe <30).
* drink cure Contraindication (500 ml/d for 21 days).
* Contraindication to any drug in the study, including a known allergy, especially magnesium.
* Uncontrolled and clinically significant heart disease, whether its origin (arrhythmias, angina, uncompensated congestive heart failure).
* Subject participating to an other clinical study interventional.
* Person deprived of liberty or under legal guardianship.
* No one in the same household who participated in this study.
* Patient refusing hospitalization.
* Persons subject to sections L1121-7 and L1121-8 of the CSP (minor, person deprived of liberty by judicial or administrative decision, person subject to a legal protection measure) or not able to communicate his consent verbally.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Actual)
Dates: Start 2021-01-22 (Actual); Primary Completion 2022-05-22 (Estimated); Study Completion 2023-05-22 (Estimated)

PRIMARY OUTCOMES:
Change in the incidence rate of the onset of clinical worsening | 12 to 14 days
  Demonstrate that the daily ingestion of 250 mL twice a day, i.e. 0.5 L of water saturated with molecular hydrogen for 21 days compared to water not enriched in hydrogen, decreases the incidence rate of the appearance of clinical worsening in patients within 12 to 14 days following a COVID-19 + diagnosis with outpatient care.
  The primary endpoint is a composite endpoint combining worsening of dyspnea, fatigue, putting on 02, hospitalizations, death occurring within 12 to 14 days of inclusion in the study.
  The worsening of dyspnea, fatigue being defined as an increase of 25% via Chalder scale for fatigue, MMRC scale for dyspnea.
  Chalder scale with 11 items (mental 7 questions yes/no and physical symptoms 4 questions yes/no) MMRC scale with 4 stades (stade 0 "no dyspnea" to 4 "strong dyspnea")

SECONDARY OUTCOMES:
Assessment of tolerance | 30 days
  Evaluate the tolerance to the treatment during the first 30 days (via a logbook of symptomatic events).
Assessment of compliance | 21 days
  Evaluate compliance with treatment by the frequency, percentage of expected intake using a logbook filled in by the patient during the 21 days of taking the treatment (at least 80% using a logbook collecting symptomatic events). Frequency and percentage will be combined to report observance.
Assessment of medium-long term dyspnea symptoms | 30 Days, 3 months, 12 months
  Evaluate in the symptoms at 30 Days, 3 months, 12 months for dyspnea via the modified MMRC Borg scale. The MMRC Borg scale contains 5 questions, stade 0 for dyspnea with strong effort and stade 4 for dyspnea with light effort.
Assessment of medium-long term fatigue symptoms | 30 Days, 3 months, 12 months
  Evaluate in the symptoms at 30 Days, 3 months, 12 months for fatigue via the Chalder scale. The Chalder scale contains 2 domains (physical and mental symptoms), with a total of 11 questions yes/no, answer yes correspond to the presence of symptom.
Assessment of oximetry symptoms | 30 Days
  Evaluate in the symptoms at 30 Days for pulse oximetry during the first 30 days. Pulse oximetry will be reported daily by the patient on the logbook (one measure/day).
Assessment of quality of life | 30 days, 3 months, 12 months
  Evaluate the quality of life via EQ5D5L scale. EQ-5D-5L is a standardized instrument developed by the EuroQol Group as a measure of health-related quality of lige that can be used in a wide range of health conditions and treatments. The EQ5D has 6 items intended to measure general health. The top 5 rate mobility, independence, daily activities, pain / discomfort, and anxiety / depression, and are rated according to 5 values : "No problem", "little problem", "moderate problem", "high problem" and "Incapacity". This results in an index score. The last item deals with perceived health on the day the questionnaire is filled in and uses a visual analogue scale from 0 (wors) to 100 (best health possible) (Visual Analog Scale Score)
Assesment of sleep quality | 30 days, 3 months, 12 months
  Evaluate the quality of sleep by PSQI scale (11 questions). The PSQI scale (Pittsburgh Sommeil Qualité Index) contains 19 questions (auto evaluation) and 5 questions for nearby. A total score of 21 points will be obtained (0 for no difficulties, 21 for major difficulties).
Assessment of care consumption | 30 days, 3 months, 12 months
  Evaluate the consumption of care via the patient notebook (hospitalizations, medical consultations).
Assessment of blind treatment | 30 days
  Evaluate the blind by CRA survey (question by phone on the potential drug group)
Assessment of COVID-19 contact cases | 30 days
  Evaluate the number of COVID-19 among contact cases per CRA survey
Assessment of risk factors | 30 days, 3 months, 12 months
  Evaluate the risk factors (age, comorbidities), physical activity, nutritional status (weight) before and after COVID-19 infection via the patient notebook. Comorbidities, physical activity, nutritional status will be combined to report risk factors.
Analysis of older patients | inclusion
  Sub group analysis on the primary outcome measure (stratification on age at inclusion > or = 70 years).
Assessment of pain | 14 days, 30 days, 3 months, 12 months
  Evaluate the pain via regular EVA score, DN4 (Douleur Neuropathique 4) Questionnaire (10 questions/4 domains) a total score will be obtain (0 no neuropathic pain, 10 major neuropathic pain).

CONTACTS AND LOCATIONS:
Overall Officials: Yoann Gaboreau, Dr, Principal Investigator — Laboratoire TIMC Equipe Themas
Locations (3):
- Timc-Imag (Umr5525 Uga-Cnrs), Grenoble, France
- Casablanca center, Casablanca, Morocco
- Public Health Center, Kamenitz, Serbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Mehta P, McAuley DF, Brown M, Sanchez E, Tattersall RS, Manson JJ; HLH Across Speciality Collaboration, UK. COVID-19: consider cytokine storm syndromes and immunosuppression. Lancet. 2020 Mar 28;395(10229):1033-1034. doi: 10.1016/S0140-6736(20)30628-0. Epub 2020 Mar 16. No abstract available. PMID 32192578
- [Background] Thompson BT, Chambers RC, Liu KD. Acute Respiratory Distress Syndrome. N Engl J Med. 2017 Aug 10;377(6):562-572. doi: 10.1056/NEJMra1608077. No abstract available. PMID 28792873
- [Background] TY - JOUR AU - Russell, Grace AU - Veal, David AU - Rehman, Mubasher AU - Adukwu, Emmanuel AU - LeBaron, Tyler AU - Hancock, John PY - 2020/06/22 SP - T1 - An Overview of SARS-CoV-2 (COVID-19) Infection and the Importance of Molecular Hydrogen as an Adjunctive Therapy DO - 10.20455/ros.2020.829 JO - Reactive Oxygen Species ER -
- [Background] Dole M, Wilson FR, Fife WP. Hyperbaric hydrogen therapy: a possible treatment for cancer. Science. 1975 Oct 10;190(4210):152-4. doi: 10.1126/science.1166304.
- [Background] Ohsawa I, Ishikawa M, Takahashi K, Watanabe M, Nishimaki K, Yamagata K, Katsura K, Katayama Y, Asoh S, Ohta S. Hydrogen acts as a therapeutic antioxidant by selectively reducing cytotoxic oxygen radicals. Nat Med. 2007 Jun;13(6):688-94. doi: 10.1038/nm1577. Epub 2007 May 7. PMID 17486089
- [Background] Itoh T, Hamada N, Terazawa R, Ito M, Ohno K, Ichihara M, Nozawa Y, Ito M. Molecular hydrogen inhibits lipopolysaccharide/interferon gamma-induced nitric oxide production through modulation of signal transduction in macrophages. Biochem Biophys Res Commun. 2011 Jul 22;411(1):143-9. doi: 10.1016/j.bbrc.2011.06.116. Epub 2011 Jun 23. PMID 21723254
- [Background] Manaenko A, Lekic T, Ma Q, Zhang JH, Tang J. Hydrogen inhalation ameliorated mast cell-mediated brain injury after intracerebral hemorrhage in mice. Crit Care Med. 2013 May;41(5):1266-75. doi: 10.1097/CCM.0b013e31827711c9. PMID 23388512
- [Background] Xie K, Yu Y, Zhang Z, Liu W, Pei Y, Xiong L, Hou L, Wang G. Hydrogen gas improves survival rate and organ damage in zymosan-induced generalized inflammation model. Shock. 2010 Nov;34(5):495-501. doi: 10.1097/SHK.0b013e3181def9aa. PMID 20351628
- [Background] Xie K, Fu W, Xing W, Li A, Chen H, Han H, Yu Y, Wang G. Combination therapy with molecular hydrogen and hyperoxia in a murine model of polymicrobial sepsis. Shock. 2012 Dec;38(6):656-63. doi: 10.1097/SHK.0b013e3182758646. PMID 23160520
- [Background] Xie K, Yu Y, Huang Y, Zheng L, Li J, Chen H, Han H, Hou L, Gong G, Wang G. Molecular hydrogen ameliorates lipopolysaccharide-induced acute lung injury in mice through reducing inflammation and apoptosis. Shock. 2012 May;37(5):548-55. doi: 10.1097/SHK.0b013e31824ddc81. PMID 22508291
- [Background] LeBaron TW, Kura B, Kalocayova B, Tribulova N, Slezak J. A New Approach for the Prevention and Treatment of Cardiovascular Disorders. Molecular Hydrogen Significantly Reduces the Effects of Oxidative Stress. Molecules. 2019 May 31;24(11):2076. doi: 10.3390/molecules24112076. PMID 31159153
- [Background] Ohta S. Molecular hydrogen as a preventive and therapeutic medical gas: initiation, development and potential of hydrogen medicine. Pharmacol Ther. 2014 Oct;144(1):1-11. doi: 10.1016/j.pharmthera.2014.04.006. Epub 2014 Apr 24. PMID 24769081
- [Background] Ono H, Nishijima Y, Adachi N, Sakamoto M, Kudo Y, Kaneko K, Nakao A, Imaoka T. A basic study on molecular hydrogen (H2) inhalation in acute cerebral ischemia patients for safety check with physiological parameters and measurement of blood H2 level. Med Gas Res. 2012 Aug 23;2(1):21. doi: 10.1186/2045-9912-2-21. PMID 22916706
- [Background] Abraini JH, Gardette-Chauffour MC, Martinez E, Rostain JC, Lemaire C. Psychophysiological reactions in humans during an open sea dive to 500 m with a hydrogen-helium-oxygen mixture. J Appl Physiol (1985). 1994 Mar;76(3):1113-8. doi: 10.1152/jappl.1994.76.3.1113. PMID 8005852
- [Background] Fontanari P, Badier M, Guillot C, Tomei C, Burnet H, Gardette B, Jammes Y. Changes in maximal performance of inspiratory and skeletal muscles during and after the 7.1-MPa Hydra 10 record human dive. Eur J Appl Physiol. 2000 Mar;81(4):325-8. doi: 10.1007/s004210050050. PMID 10664092
- [Background] Zhou ZQ, Zhong CH, Su ZQ, Li XY, Chen Y, Chen XB, Tang CL, Zhou LQ, Li SY. Breathing Hydrogen-Oxygen Mixture Decreases Inspiratory Effort in Patients with Tracheal Stenosis. Respiration. 2019;97(1):42-51. doi: 10.1159/000492031. Epub 2018 Sep 18. PMID 30227423
- [Background] Hu Y, Sun J, Dai Z, Deng H, Li X, Huang Q, Wu Y, Sun L, Xu Y. Prevalence and severity of corona virus disease 2019 (COVID-19): A systematic review and meta-analysis. J Clin Virol. 2020 Jun;127:104371. doi: 10.1016/j.jcv.2020.104371. Epub 2020 Apr 14. PMID 32315817
- [Background] Verity R, Okell LC, Dorigatti I, Winskill P, Whittaker C, Imai N, Cuomo-Dannenburg G, Thompson H, Walker PGT, Fu H, Dighe A, Griffin JT, Baguelin M, Bhatia S, Boonyasiri A, Cori A, Cucunuba Z, FitzJohn R, Gaythorpe K, Green W, Hamlet A, Hinsley W, Laydon D, Nedjati-Gilani G, Riley S, van Elsland S, Volz E, Wang H, Wang Y, Xi X, Donnelly CA, Ghani AC, Ferguson NM. Estimates of the severity of coronavirus disease 2019: a model-based analysis. Lancet Infect Dis. 2020 Jun;20(6):669-677. doi: 10.1016/S1473-3099(20)30243-7. Epub 2020 Mar 30. PMID 32240634
- [Background] Chow SC, Shao J, Wang H. A note on sample size calculation for mean comparisons based on noncentral t-statistics. J Biopharm Stat. 2002 Nov;12(4):441-56. doi: 10.1081/BIP-120016229. PMID 12477068
- [Background] LeBaron, T. W., McCullough M. L. and Ruppman Sr K. H., A novel functional beverage for COVID-19 and other conditions: Hypothesis and preliminary data, increased blood flow, and wound healing, Journal of Translational Science, 6(2020), pp 1-6, doi: 10.15761/JTS.1000380
- [Background] Guan WJ, Wei CH, Chen AL, Sun XC, Guo GY, Zou X, Shi JD, Lai PZ, Zheng ZG, Zhong NS. Hydrogen/oxygen mixed gas inhalation improves disease severity and dyspnea in patients with Coronavirus disease 2019 in a recent multicenter, open-label clinical trial. J Thorac Dis. 2020 Jun;12(6):3448-3452. doi: 10.21037/jtd-2020-057. No abstract available. PMID 32642277
- [Background] Haute Autorité de Santé. Réponses rapides dans le cadre de la Covid-19 - Prise en charge de premier recours des patients suspectés de Covid-19. Paris,18 juin 2020. Mise à jour en nov. 2020
- See also: High Council of Public Health. Opinion of 29 October 2020 on the updating of the list of risk factors for the severe form of COVID-19 — http://www.hcsp.fr/Explore.cgi/AvisRapportsDomaine?clefr=942
- See also: High Authority of Health. Rapid responses in the context of Covid-19 - Primary care of patients suspected of Covid-19. Paris, June 18, 2020. Updated in Nov 2020 — http://www.has-sante.fr/upload/docs/application/pdf/2020-04/reponse_rapide_covid19_malchron.pdf